CLINICAL TRIAL: NCT05084989
Title: A Randomized, Blinded, Two-part, Phase II Trial to Evaluate the Safety and Immunogenicity of the Recombinant Two-component COVID-19 Vaccine (CHO Cell) in Adults 18 Years and Older
Brief Title: Safety, and Immunogenicity Study of the Recombinant Two-component COVID-19 Vaccine (CHO Cell)
Acronym: ReCOV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu Rec-Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: REC611C301
Record Dates: First submitted 2021-10-14; First posted 2021-10-20 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — RNA, Messenger

STUDY DESIGN:
Intervention Model Description: Part1: 2 arms Part2: 2 arms
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part1: double blinded Part2: observer-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part1: Recombinant two-component COVID-19 vaccine (CHO cell) (Experimental): Antigen: NTD-RBD-foldon protein, sodium dihydrogen phosphate, disodium hydrogen phosphate, sucrose, glycine, polysorbate 80 Adjuvant (BFA03): squalene, alpha-tocopherol, polysorbate 80, sodium chloride, potassium chloride, disodium hydrogen phosphate, potassium dihydrogen phosphate
  Interventions: Biological: Part1:Recombinant two-component COVID-19 vaccine (CHO cell)
- Part1: Placebo control (Placebo Comparator): Antigen: sodium dihydrogen phosphate, disodium hydrogen phosphate, sucrose, glycine, polysorbate 80 Adjuvant (BFA03): squalene, alpha-tocopherol, polysorbate 80, sodium chloride, potassium chloride, disodium hydrogen phosphate, potassium dihydrogen phosphate
  Interventions: Biological: Part1: Placebo
- Part2: Recombinant two-component COVID-19 vaccine (CHO cell) (Experimental): (Lot# HA202107009 and Lot# TC202205002) Recombinant two-component COVID-19 vaccine (CHO cell) Antigen: NTD-RBD-foldon protein, sodium dihydrogen phosphate, disodium hydrogen phosphate, sucrose, glycine, polysorbate 80 Adjuvant (BFA03): squalene, alpha-tocopherol, polysorbate 80, sodium chloride, potassium chloride, disodium hydrogen phosphate, potassium dihydrogen phosphate
  Interventions: Biological: Part2: Recombinant two-component COVID-19 vaccine (CHO cell)
- Part2: COMIRNATY® COVID-19 Vaccine, mRNA (Active Comparator): Antigen: nucleoside-modified messenger RNA (mRNA) encoding the viral Spike (S) glycoprotein of SARS-CoV-2, called tozinameran.
  Others: ((4-hydroxybutyl) azanediyl) bis (hexane-6,1-diyl) bis (2-hexyldecanoate), 2-[(polyethylene glycol)-2000]-N, N-ditetradecylacetamide, 1,2-distearoyl-sn-glycero-3-phosphocholine, and cholesterol, potassium chloride, potassium dihydrogen phosphate, sodium chloride, disodium phosphate dihydrate, sucrose.
  Interventions: Biological: Part2: COVID-19 Vaccine, mRNA

INTERVENTIONS:
Biological: Part1:Recombinant two-component COVID-19 vaccine (CHO cell) — 2 doses. Before reconstitution:Lyophilized powder for reconstitution in single-use vials; After reconstitution with BFA03 adjuvant: Milk-white solution with no visible foreign matter; Unite Does Strengths: 40ug/vial; Does Volume: 0.5ml/dose Routine of administration: Intramuscular (IM) injection
  Other Names: Part1: ReCOV
  Arms: Part1: Recombinant two-component COVID-19 vaccine (CHO cell)
Biological: Part1: Placebo — 2 doses. Before reconstitution: Lyophilized powder for reconstitution in single-use vials; After reconstitution with BFA03 adjuvant: Milk-white solution with no visible foreign matter; Unite Does Strengths: Not Applicable; Does Volume: 0.5ml/dose; Routine of administration: IM injection;
  Arms: Part1: Placebo control
Biological: Part2: Recombinant two-component COVID-19 vaccine (CHO cell) — 1 dose.Before reconstitution:Lyophilized powder for reconstitution in single-use vials; After reconstitution with BFA03 adjuvant: Milk-white solution with no visible foreign matter; Unite Does Strengths: 40ug/vial; Does Volume: 0.5ml/dose Routine of administrati
  Other Names: Part2: ReCOV
  Arms: Part2: Recombinant two-component COVID-19 vaccine (CHO cell)
Biological: Part2: COVID-19 Vaccine, mRNA — 1 dose. Intramuscular injection, 30 μg/0.3 mL.
  Other Names: Part2: COMIRNATY®
  Arms: Part2: COMIRNATY® COVID-19 Vaccine, mRNA

SUMMARY:
Part 1: Primary Vaccination in Adults Part 1 will evaluate the safety and immunogenicity of the recombinant two component COVID-19 vaccine (CHO cell) (ReCOV for short) in adults aged 18 years and older, when administered as 2 intramuscular doses, 21 days apart.

Part 2: Booster Vaccination in Adults Part 2 will evaluate the immunogenicity and safety and of one booster dose of ReCOV in adult participants who have received primary vaccination with 2 doses of an inactivated COVID-19 vaccine (CoronaVac®). COMIRNATY®, an mRNA COVID-19 vaccine will be used as the active control.

DETAILED DESCRIPTION:
Part 1: Primary Vaccination in Adults Around 340 participants aged 18 years and older who do not have known COVID-19 or COVID-19 vaccination history will be randomized into ReCOV group (40 μg) or placebo group in a ratio of 2:1. Accordingly, around 227 participants will receive 40 μg ReCOV and 113 participants will receive matching placebo, respectively. Participants will be stratified by age (18~59 years, ≥60 years) and status of SARS-CoV-2 antibody at baseline.

After randomization, participants will enter into a double-blinded period (until all participants complete V6) and an open-label long-term follow-up period (after all participants complete V6 until end of the study).

After all participants complete the visit at 7 days after the 2nd vaccination, the safety and reactogenicity data will be summarized by an independent statistic group, while the sponsor, investigators and all study participants will be kept blinded. The safety summary will be submitted to DSMB for review and recommendation on the initiation of Part 2.

The primary analysis of Part 1 is planned after all participants complete the Visit 6 (V3 + 28 days, +7 days) and are unblinded, to evaluate the safety and immunogenicity during the double-blinded period.

The final analysis of Part 1 will be conducted after all participants of the ReCOV group complete the follow-up visit at 6 months after the 2nd vaccination, to evaluate the safety and immunogenicity during this study stage.

Part 2: Booster Vaccination in Adults This study part will enroll participants who have received primary vaccination by an inactivated COVID-19 vaccine (CoronaVac®) within 3 to 12 months (90~365 days). The mRNA COVID-19 vaccine, COMIRNATY ®, will be used as the active control. The immunogenicity induced by the booster vaccination of ReCOV (commercial batch, Lot# TC202205002) will be compared with that of COMIRNATY®. In addition, the immunogenicity of one dose booster of commercial batch ReCOV (Lot# TC202205002) will be compared with that of pilot batch ReCOV (Lot# HA202107009).

About 600 participants will be enrolled into the study. Eligible participants will be 1:1:1 randomized to receive 20 μg ReCOV (Lot# HA202107009), 20 μg ReCOV (Lot# TC202205002), or 30 μg COMIRNATY®, stratified by age (18~59 years, ≥60 years) and the duration since the last primary vaccination (90~180 days, 181~365 days).

All participants will be followed up for safety and reactogenicity. Participants will be observed for 30 minutes at study site after the vaccination. Before leaving the study site, participants will be given participant diaries to record solicited AEs within 7 days after dosing, and unsolicited AEs within 28 days after dosing. The occurrence of SAEs and AESIs will also be monitored till 6 months after the study vaccination.

The interim analysis is planned after all participants complete the Visit 5 at 28 days after the dosing, to evaluate the immunogenicity and safety within this period.

The final analysis will be conducted after all participants complete the follow-up visit at 6 months post the booster vaccination, to evaluate the immunogenicity and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years and older.
2. All participants are able and willing to comply with all study requirements.
3. Willing to allow investigators to discuss the medical history with his/her general practitioner/personal doctors and access all medical records which are relevant to study procedures.
4. Healthy participants, or participants with stable medical condition who have a pre-existing medical condition that does not meet any exclusion criteria. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.
5. For Part 1, participants should have not received any COVID-19 vaccine before the screening.

   For Part 2, participants should have received complete 2-dose primary vaccination with an inactivated COVID-19 vaccine (CoronaVac®), 90~365 days (included) prior to the study vaccination.
6. Provide written informed consent form (ICF) prior to study enrollment.

Exclusion Criteria

1. Laboratory confirmed SARS-CoV-2 infection, defined by RT-PCR assay.
2. Medical history of severe acute respiratory syndrome (SARS), middle east respiratory syndrome (MERS) and COVID-19 within 12 months prior to the randomization.
3. Fever (oral temperature ≥ 37.5°C / axillary temperature ≥ 37.3°C) on the day of vaccination or within recent 72 hours.
4. History of severe allergic disease or reactions likely to be exacerbated by any component of ReCOV or the control vaccine, such as allergic shock, allergic laryngeal edema, allergic purpura, thrombocytopaenic purpura, local hypersensitive necrosis reaction (Arthus reaction), or prior history of serious adverse reaction to any vaccine or drug, such as allergy, urticaria eczema, dyspnea, and angioneurotic edema.
5. Have malignant tumor (except for skin basal cell carcinoma or carcinoma uterine cervix in situ) and immune disease (e.g., human immunodeficiency virus [HIV] infection, systemic lupus erythematosus, rheumatoid arthritis, asplenia or splenectomy, and other immune disease that may influence immune response at investigator's discretion).
6. Have other severe and/or uncontrolled conditions, including but not limited to, acute infectious disease, cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, hematology disease, endocrine disorder, psychiatric condition and neurological illness. Mild/moderate well-controlled comorbidities are allowed to participate as deemed appropriate by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 948 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2022-08-18 (Actual); Study Completion 2023-02-09 (Actual)

PRIMARY OUTCOMES:
Part1, Primary Safety | Day 7 after first dose and up to Day 28 after second dose
  Number of Participants with AEs
Part1, Primary immunogenicity | 14 days after 2 doses vaccination
  To evaluate SARS-CoV-2 Specific Neutralizing Antibody
Part2, Primary immunogenicity | 14 days after 2 doses vaccination
  To evaluate SARS-CoV-2 Specific Neutralizing Antibody

SECONDARY OUTCOMES:
Part1, Immunogenicity | 14 days, 3 months and 6 months after 2 doses vaccination
  To evaluate other immunogenicity variables of ReCOV in adults aged 18 years and older.
Part2, safety and reactogenicity | 7 days, 28days and 6 months after the booster vaccination
  The occurrence of AEs

CONTACTS AND LOCATIONS:
Overall Officials: fanyue Meng, Principal Investigator — cdc jiangsu
Locations (1):
- The Health Centrum, Roxas City, Philippines

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available

REFERENCES:
- [Derived] Balgos A, Hannawi S, Chen WL, Abuquta A, Safeldin L, Hassan A, Alamadi A, Tirador L, Jaen AM, Villalobos RE, Mo C, Yue ZJ, Ma Y, Wang QS, Wen RD, Yao Z, Yu JP, Yao WR, Zhang JH, Hong KX, Liu Y, Li JX. Immunogenicity and safety of boosting with a recombinant two-component SARS-CoV-2 vaccine: two randomized, parallel-controlled, phase 2 studies. Expert Rev Vaccines. 2024 Jan-Dec;23(1):419-431. doi: 10.1080/14760584.2024.2334423. Epub 2024 Apr 2. PMID 38529685
- [Derived] Wynne C, Balgos A, Li J, Hamilton P, Tirador L, Jaen AM, Mo C, Yue Z, Ma Y, Wang Q, Wen R, Yao Z, Yu J, Yao W, Zhang J, Zheng H, Hong K, Zhu F, Liu Y. Safety and Immunogenicity of a Recombinant Two-Component SARS-CoV-2 Protein Vaccine: Randomized, Double-Blind, Placebo-Controlled Phase I and Phase II Studies. Infect Dis Ther. 2024 Jan;13(1):57-78. doi: 10.1007/s40121-023-00896-w. Epub 2023 Dec 16. PMID 38103161